CLINICAL TRIAL: NCT00103766
Title: Randomized Comparison of Two Dose and Frequency Regimens of Alteplase for Treatment of Empyema and Complicated Parapneumonic Effusion
Brief Title: Alteplase for Treatment of Empyema and Complicated Parapneumonic Effusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: O'Brien, Jeana D., MD, FACP, FCCP (Individual)
Collaborators: Genentech, Inc. (Industry); Scott and White Hospital & Clinic (Other); Scott, Sherwood and Brindley Foundation (Other); Texas A&M University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8736
Record Dates: First submitted 2005-02-14; First posted 2005-02-15 (Estimated); Last update posted 2006-08-01 (Estimated); Status verified 2006-07

CONDITIONS: Empyema; Pleural Effusion
Keywords: Alteplase; Empyema; Complicated Parapneumonic Effusion
MeSH Terms: conditions — Empyema; Pleural Effusion | interventions — Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Alteplase

SUMMARY:
The purpose of this study is to assess the benefit to patients with empyema or complicated parapneumonic effusion (CPE) using a daily versus twice daily Alteplase regimen of two different dose strategies compared with saline placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled pilot study. Patients with empyema and complicated parapneumonic effusion who are felt to require fibrinolytic therapy will be considered for study enrollment. Enrolled patients will be randomized to one of five potential treatment arms (saline placebo, 4 mg once daily, 4 mg twice daily, 10 mg once daily, or 10 mg twice daily) in a double-blinded manner.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Age greater or equal to 18 yrs
* Presence of empyema or CPE

Exclusion Criteria:

* Active internal bleeding
* Pregnancy
* Prior enrollment in this study
* Platelet count less than 100,000/mm3
* Use of warfarin sodium if INR is greater than 1.7
* Use of heparin unless the PTT is less than 1.5 times baseline normal
* Known neurological disorders
* Current or pre-existing bleeding dyscrasia
* Known allergy to Alteplase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2004-10

PRIMARY OUTCOMES:
Need for surgical intervention via thoracostomy or open decortication as a result of conservative therapy.

SECONDARY OUTCOMES:
Mortality
Hospital length of stay
Daily chest tube drainage
Radiographic improvement

CONTACTS AND LOCATIONS:
Overall Officials: Jeana D O'Brien, MD, FACP, FCCP, Principal Investigator — Scott and White Memorial Hospital and Scott, Sherwood and Brindley Foundation
Locations (1):
- Scott and White Memorial Hospital & Clinic, Temple, Texas, United States